CLINICAL TRIAL: NCT03116880
Title: In Vivo Evaluation of Image Registration Techniques During Endovascular Repair
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 2016/533
Record Dates: First submitted 2017-04-11; First posted 2017-04-17 (Actual); Last update posted 2018-09-05 (Actual); Status verified 2018-09

CONDITIONS: Aortic Aneurysm, Abdominal
Keywords: Aorta, Abdominal/surgery; Endovascular Procedures
MeSH Terms: conditions — Aortic Aneurysm, Abdominal | interventions — Endovascular Aneurysm Repair

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Image registration
  Interventions: Procedure: Endovascular aortic repair

INTERVENTIONS:
Procedure: Endovascular aortic repair — Endovascular aortic repair

SUMMARY:
Fluoroscopy is traditionally used for guidance of endovascular aortic repair (EVAR). In order to minimize exposure to radiation and nephrotoxic contrast medium, it is possible to generate a navigation road map by registering the intraoperative images with preoperative computed tomography angiograph (CTA). In modern hybrid operating rooms, several commercial solutions for this exists today (e.g. Siemens Syngo iPilot, Phillips Vesselnavigator). In order to register (fuse) the preoperative and intraoperative imaging to each other, a registration algorithm has to be applied. Sufficient accuracy of this algorithm is crucial, for if it fails the road map cannot be used for intraoperative navigation. The purpose of this study is therefore to evaluate two different 3D registration algorithms with regard to registration accuracy.

DETAILED DESCRIPTION:
Two different registration algorithms will be tested:

1. registration algorithm - centerline registration algorithm (Sintef, Trondheim) A catheter equipped with a position sensor records the travelled path of the instrument, which is assumed to be close to the centerline of the aorta. From the preoperative computer tomography scan (CT) the aorta is segmented and vessel centerline is extracted. The centerline from the position sensor recordings is registered to the extracted centerline of the preoperative CT.
2. 3D-3D registration algorithm (Syngo iPilot, Siemens Medical Solutions, Munich). Intraoperative cone-beam-CT (CBCT) is registered to the preoperative CT

ELIGIBILITY:
Inclusion Criteria:

* infrarenal or juxtarenal abdominal aortic aneurysm
* undergoing EVAR
* informed consent

Exclusion Criteria:

* under 18 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients undergoing endovascular aortic repair at St. Olav Hospital, Trondheim, Norway
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2017-04-19 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Registration accuracy of registration algorithms | Immediately
  Measure the 3D spread between defined points (registration plate, bony landmarks at vertebrae, vessels if visable)

CONTACTS AND LOCATIONS:
Overall Officials: Øystein Risa, Study Director — Norwegian University of Science and Technology, Department of Circulation and Medical Imaging
Locations (1):
- St. Olavs hospital, Trondheim, Norway

IPD SHARING:
Plan to Share IPD: Undecided